CLINICAL TRIAL: NCT01487551
Title: An Open-Label Study to Evaluate Biomarkers and Safety in Systemic Sclerosis Patients Treated With ABR-215757 (Paquinimod)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Active Biotech AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11575705; 2011-001667-44 (EudraCT Number)
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2014-08-27 (Estimated); Status verified 2014-08

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis; Biomarkers
MeSH Terms: conditions — Scleroderma, Systemic | interventions — paquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- paquinimod (Experimental)
  Interventions: Drug: paquinimod

INTERVENTIONS:
Drug: paquinimod — Hard gelatine capsules 3.0 mg/day for 8 weeks

SUMMARY:
The primary objective is to study changes in disease related biomarkers in patients with progressive SSc during treatment with ABR-215757.

The secondary objectives are to assess the safety and tolerability of ABR-215757,to assess disease activity and quality of life (QoL)during treatment with ABR-215757 and to assess the plasma levels of ABR-215757 during the study.

DETAILED DESCRIPTION:
This is an open label single arm Phase II study in patients with progressive SSc. Patients will be treated with ABR-215757 for 8 weeks. Assessment of biomarkers, disease activity and safety parameters will be performed during treatment. Patients will be offered to continue in an open label extension.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing the informed consent form
2. Clinical Diagnosis of SSc according to ACR criteria
3. Progressive SSc fulfilling at least one of the following:

   * STPR (Skin Thickness Progression Rate) ≥ 40, calculated as the mRSS at screening divided by time (in years) since the start of skin involvement. as reported by the patient (Denton 2007)
   * Worsening of mRSS within the last 6 months as judged by the physician together with the patient, with involvement of at least two new anatomical sites as defined in the mRSS score (e.g. upper arm and thorax) or progression by at least two points in at least two anatomical sites as defined by the mRSS
4. Presence of SSc skin lesions on one or both forearms
5. Modified Rodnan Skin score (mRSS) ≥16 at baseline
6. ANA-positive

Exclusion Criteria:

1. Ongoing Severe SSc manifestations, such as pulmonary arterial hypertension (PAH) with dyspnea NYHA III or more, scleroderma renal crisis
2. Vital capacity < 60% as measured within 6 months prior to the first dose of study medication
3. GFR < 30% of normal measured within 6 months prior to the first dose of study medication
4. Treatment with Rituximab within 12 months or other biologic agent within 6 months, Mycophenolate mofetil (MMF) or Cyclophosphamide within 6 months, Methotrexate, Azathioprine or other immunosuppressants within 3 months prior to the first dose of study medication
5. History of myocardial infarction or current uncontrolled angina, severe uncontrolled ventricular arrhythmias, symptomatic congestive heart failure, unstable angina pectoris, or electrocardiographic evidence of acute ischemia.
6. Marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval >450 milliseconds
7. History of additional risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome)
8. Treatment with concomitant medications that prolong the QT interval.
9. History of, or current ischemic CNS disease
10. Current malignancy. A 5-year cancer-free period is required with the exception of skin basal or squamous cell carcinoma or cervical cancer in situ that has been excised
11. Current severe infection
12. Known positive serology for HIV or active or latent hepatitis infection.
13. Treatment with endothelin receptor antagonist within 6 weeks prior to the first dose of study medication
14. Drug abuse
15. Major surgery within 3 weeks prior to study entry
16. Known or suspected hypersensitivity to ABR-215757 or excipients
17. Female patient of child-bearing potential who is not using a medically accepted safe method of contraception. All female patients of child-bearing potential must have a negative urine pregnancy test at the Screening and Baseline Visits. As interaction studies between ABR-215757 and hormonal contraceptives have not yet been performed, women using hormonal contraceptives such as the contraceptive pill, must also use a complementary contraceptive device, i.e. barrier method, during the treatment period and for at least 1 month thereafter
18. Female patient of child-bearing potential who is pregnant or lactating.
19. Simultaneous participation or participation within 4 months or 5 half lives (whichever is longer) prior to study entry in any other study involving investigational drugs or other experimental therapy.
20. Other significant, unstable medical disease not related to SSc that in the investigator's opinion would confound the study result or put the patient at risk
21. Patients likely to receive oral or intravenous steroids or immunosuppressant for other non-SSc condition during the study duration, as this will confound the study result.
22. Vaccination within 4 weeks prior to the first dose of study medication. Study Drug(s): ABR-215757

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Biomarkers | Assessment of biomarkers will be performed at baseline, after 2, 4, and 8 weeks of treatment.
  Changes in SSc disease activity related biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Roger Hesselstrand, MD, Principal Investigator — Dept of Rheumatology, University Hospital in Lund, Sweden
Locations (6):
- Germany (3):
  - Berlin
  - Cologne
  - Erlangen
- Sweden (2):
  - Gothenburg
  - Lund
- Zurich, Switzerland

REFERENCES:
- [Derived] Hesselstrand R, Distler JHW, Riemekasten G, Wuttge DM, Torngren M, Nyhlen HC, Andersson F, Eriksson H, Sparre B, Tuvesson H, Distler O. An open-label study to evaluate biomarkers and safety in systemic sclerosis patients treated with paquinimod. Arthritis Res Ther. 2021 Jul 31;23(1):204. doi: 10.1186/s13075-021-02573-0. PMID 34330322